CLINICAL TRIAL: NCT05449223
Title: Evaluation of Reliability and Validity of Urdu Version of the Frenchay Activities Index in Pakistani Geriatric Population
Brief Title: Urdu Version of Frenchay Activities Index: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00241
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Activity, Motor
Keywords: Frenchay Activities Index; Urdu Version; Activities of Daily Living; Validity; Reliability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we will observe the reliability and validity of frenchay activities index and barthel index in urdu language in geriatric population of Pakistan.

DETAILED DESCRIPTION:
The aim of study is to translate and culturally adapt Frenchay Activities Index and Bathel Index into Urdu language and secondly to investigate the reliability and validity of Frenchay Activities Index and Barthel Index in geriatric population of Pakistan. This study will be cross sectional survey study in which convenience sampling technique will be used.

The results of study will help to know the validity and reliability of Frenchay Activities Index and Barthel Index in Urdu version with Activities of Daily Livings impairments in geriatric population of Pakistan. The reliability of the questionnaire will be checked through internal consistency and test-retest methods. internal consistency will be analyzed with Cronbach's alpha value. Test-retest reliability will be assessed using an intra-class correlation coefficient with 75 patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and older
* be able to read Urdu
* be living in Pakistan for more than 5 years
* have minimal cognitive impairment with Mini-Mental State Examination
* have no significant muscle, joint, or neurologic conditions such as stroke, or Parkinson's disease.

Exclusion Criteria:

* inability to understand to follow the instructions of Frenchay Activities Index and Barthel Index
* experience with the Frenchay Activities Index and Bathel Index in the last 6 months
* acute illness or fracture in the lower extremities

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly people, especially those of the advanced ages having issue in performing in activities of daily living
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Frenchay activities index | 12th Week
  Frenchay Activities Index is used to measure performance in activities of daily living. It contains 15 items on common daily activities such as preparing a meal, washing the dishes, housekeeping, shopping, hobbies, going out, and work. The patient is asked whether or not he/she did the activities for the past 3-6 months. The scores are from 1 (never) to 4 (normal frequency) with a total score range from 15 to 60. A lower score means a lower level of functioning.
Barthel Index | 12th Week
  Barthel Index is used to measure performance in activities of daily living. The Barthel Index contains 10 items on sphincter control, grooming, toilet use, eating, transfer, and mobility compromising one dimension on the need for help. The score differs per item and the total score ranges from 0 (totally dependent) to 20 (independent).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No